CLINICAL TRIAL: NCT05299450
Title: Pre-conception Interventions to Reduce Blood Pressure Before Pregnancy
Acronym: CONCEIVE 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274808
Record Dates: First submitted 2022-02-07; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Pre-conception; Hypertension; Exercise; Beetroot; Wearable
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise intervention (Experimental): 12 week personalised exercise intervention with personal trainer and gym membership, fitbit
  Interventions: Behavioral: Exercise
- Beetroot juice (Experimental): 12 weeks daily Beet It (beetroot shots) containing nitrate, fitbit
  Interventions: Dietary Supplement: Beet It shots
- Exercise and Beetroot (Experimental): 12 week personalised exercise intervention with personal trainer and gym membership and daily Beet It (beetroot shots) containing nitrate, fitbit
  Interventions: Dietary Supplement: Beet It shots; Behavioral: Exercise
- Control group (Active Comparator): No intervention, fitbit
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: Beet It shots — In addition to the procedures for the control group, women will be supplied with 84 Beet-It shots which they will be asked to take every morning with breakfast for 12 weeks. Women below 60kg will be advised to take a proportion of the 'shot' in order to comply with European Commission Accepted Daily Intake for nitrate, the active ingredient, of 0-5mg/kg. https://www.beet-it.com/product/beet-it-sport-shot/
  Arms: Beetroot juice; Exercise and Beetroot
Behavioral: Exercise — In addition to the procedures for the control group, women will be supplied with gym membership for 12 weeks, 2 initial personal training sessions to design a personal exercise program followed by monthly personal training sessions.
  Arms: Exercise and Beetroot; Exercise intervention
Other: Control group — Women will be supplied with a wearable device to measure physical activity, weighing scales and a home blood pressure monitor. They will be asked to record minutes of physical activity, exercise undertaken, resting blood pressure, resting heart rate and weight daily for 12 weeks.
  Arms: Control group

SUMMARY:
The study proposes to evaluate the feasibility of a preconception intervention comprising two proven interventions for reducing blood pressure; Beetroot juice; a source of dietary nitrate which reduces BP by 8/4mmHg after 4 weeks(6); Personalised resistance and endurance exercise programme (as per CMO recommendations) which reduces BP by ~10/5mm Hg over 8-12 weeks (7).

DETAILED DESCRIPTION:
A feasibility study will be conducted for a randomised, controlled trial of preconception interventions.

The study will advertise using posters, social media and on departmental emails at Imperial College Healthcare NHS Trust or Imperial College for women aged 18-45 planning a pregnancy at any time in the future.

The study will randomise women to 1 of 4 arms Arm 1: Exercise intervention for weeks 1-12 Arm 2: Beetroot juice for weeks 1-12 Arm 3. Exercise and Beetroot juice for weeks 1-12 Arm 4: Control group

Women will be provided with daily Beetroot juice shots (as per study arm), membership to an Everybody Active centre close to their home, personal training sessions to tailor an exercise program to them (2 initial sessions then monthly), a wearable to track their physical activity and a home BP monitor.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* considering pregnancy at some time in the future
* no health contra-indications to moderate-vigorous exercise
* employed by ICHT NHS Trust or Imperial College.

Exclusion Criteria:

* Currently pregnant
* planning pregnancy during the study period, or becoming pregnant during the study period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence to intervention | Over 12 week study period
  >/= mean150 minutes/week physical acitvity recorded by Fitbit;
Adherence to intervention | Over 12 week study period
  Percent of supplied beetroot shots consumed

SECONDARY OUTCOMES:
Effect of interventions on physical activity | Week 12
  Change in minutes/week of physical activity recorded by FitBit from minutes/week of physical activity in week 1 to minutes/week of physical activity in week 12
Effect of interventions on cardiac output | Week 12
  Change in cardiac output in l/min from initial visit to final visit at week 12
Effect of interventions on total peripheral resistance | Week 12
  Change in total peripheral resistance in dyn·s/cm5 from from initial visit to final visit at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Edward WS Mullins, PhD, Principal Investigator — Imperial College Healthcare NHS Trust; Cristoph C Lees, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Available on application to PI, however this was a feasibility study